CLINICAL TRIAL: NCT02039622
Title: Cardiovascular Toxicity Induced by Antitumoral Drugs: Risk Assessment and Early Diagnosis. CARDIOTOX Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Other Study IDs: GECAME-2010-01
Record Dates: First submitted 2014-01-10; First posted 2014-01-17 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Cardiovascular Toxicity Induced by Antitumoral Drugs

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patient under study condition: Patient under study condition

SUMMARY:
The study is multicenter, post-authorization, observational and ambispective

DETAILED DESCRIPTION:
Cardiovascular toxicity produced by antitumoral drugs has a considerable impact in life wellness and prognosis of cancer patients, which can imply the suspension of the desired antitumoral treatment or even risk the patient´s life. The development of a risk score for these patients, as well as specific methodology for early detection of cardiotoxicity would therefore be a great outcome to trigger new strategies for the monitoring of these patients. Currently there is a lack of a clinical score to predict cardiotoxicity risk. Therefore, there is an urgent need to identify new myocardial injury biomarkers and novel imaging parameters for measuring ventricular function that would increase the sensitivity of the traditional methods used for the early detection of cardiotoxicity.

The objectives of the present study are the following:

* Identify the factors related with cardiotoxicity risk produced by antitumoral drugs.
* Assess the utility of clinical, biological and functional parameters for the early detection of cardiotoxicity produced by antitumoral drugs.

The study is a multicenter one, observational and ambispective. We will include all the patients assessed by the Oncology and Haematology Departments in each participant hospital that are about to initiate or are undergoing chemotherapy with any of the drugs specified in the study protocol. Patients will be monitorized during the treatment, undergoing an echocardiography study and a blood sample collection in each clinical timepoint. All these parameters will hopefully shed some light for the development of a clinical risk score as well as identifying new early biomarkers for cardiotoxicity.

The initial follow-up in this phase of the study will be 2 years

ELIGIBILITY:
Inclusion Criteria:

* Patients> 18 years with indicated antitumor chemotherapy.
* Estimated survival ≥ 6 months
* No oxygen dependence
* No contraindication for taking the study target antitumor agents.
* No exclusion of patients with risk factors or previous heart disease.
* No exclusion of patients with previous cancer, previous antitumor treatment, current antitumor treatment, previous or current radiotherapy.
* No exclusion of patients with previous cardiovascular toxicity

Exclusion Criteria:

* No exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A case is defined as a patient on treatment (started or programmed, regardless of previous treatments or prior radiotherapy) with the following target antineoplastic agents:
  * Alkylating agents
  * Antimicrotubule agents
  * Vinca alkaloids
  * Monoclonal Antibodies
  * Antimetabolites
  * Anthracyclines
  * Angiogenesis inhibitors
  * Interleukins
  * Small molecule tyrosine kinase inhibitors
  * Other antineoplastic agents
Sampling Method: Non-Probability Sample
Enrollment: 3400 (Estimated)
Dates: Start 2011-07; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in CARDIOTOXICITY DEVELOPMENT RISK SCORE | 21 days, 3 months, 6 months, 1 year, 1.5 years and 2 years
  Risk of cardiovascular toxicity by antitumoral agents is multifactorial.
  * Clinical heart failure
  * Asymptomatic ventricular dysfunction
  * Elevated biomarkers
  * Severe arrhythmias
  * Myocardial ischemia
  * Other cardiac events
change in EARLY DETECTION OF CARDIOTOXICITY | 21 days, 3 months, 6 months, 1 year, 1.5 years and 2 years
  Early recognition of cardiotoxicity can help determine whether to continue treatment with a particular type of drug and set up preventive treatments.
  * Demographic variables for study inclusion
  * Clinical symptoms of cardiac disease
  * EKG
  * Transthoracic echocardiogram
  * Biological markers: Troponin I (cTnI), NTproBNP
  * Oncological variables: Diagnosis and cancer location, Drugs

SECONDARY OUTCOMES:
Incidence of cardiovascular toxicity in its different forms | 2 years
  Cardiotoxicity severity:
  * Mild: asymptomatic, no hospitalization needed
  * Severe: requires admission or specific treatment initiated for this reason
Incidence of cardiovascular toxicity in relation to the cumulative dose | 21 days, 3 months, 6 months, 1 year, 1.5 years and 2 years
  * Heart failure
  * Asymptomatic ventricular dysfunction
  * Myocardial Ischemia
  * Severe arrhythmias
  * Other cardiac pathology
•Incidence of cardiovascular toxicity in relation to the kind of antitumor agent | 21 days, 3 months, 6 months, 1 year, 1.5 years and 2 years
  * Heart failure
  * Asymptomatic ventricular dysfunction
  * Myocardial Ischemia
  * Severe arrhythmias
  * Other cardiac pathology
•Analyze the sensitivity and specificity of EKG changes regarding new changes in biomarkers, clinical and echocardiographic parameters | 21 days, 3 months, 6 months, 1 year, 1.5 years and 2 years
  - EKG
Analyze whether alterations of biological markers predate clinical, echocardiographic and functional parameters | 21 days, 3 months, 6 months, 1 year, 1.5 years and 2 years
  * Troponin I
  * NT-proBNP
Compare the effectiveness of early identification of cardiovascular toxicity of high-sensitivity troponin (troponin T) compared to a conventional troponin | 21 days, 3 months, 6 months, 1 year, 1.5 years and 2 years
  * Troponin I (cTn I)
  * Troponin Thigh sensitivity (cTnhs)
Define the sensitivity and specificity of the left ventricle ejection fraction in the detection of cardiovascular toxicity | 21 days, 3 months, 6 months, 1 year, 1.5 years and 2 years
  * Telediastolic volume left ventricle
  * Telesystolic volume right ventricle
  * Ejection fraction left ventricle
  * Size of left atrium
  * Size right atrium
  * Mitral valve disease
  * Tricuspid valve disease
  * Pericardial overflow
• Define the sensitivity and specificity of new ventricular function parameters in cardiovascular toxicity screening. | 21 days, 3 months, 6 months, 1 year, 1.5 years and 2 years
  - Longitudinal global strain
Economic analysis derived from the diagnostic strategy with biomarkers versus echocardiography. | 2 years
  Economic analysis comparing efficacy of biomarkers versus echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Lopez-Sendon, Principal Investigator — La Paz University Hospital- Chief of Cardiology Department
Locations (1):
- La pAz University Hospital, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Caro-Codon J, Lopez-Fernandez T, Alvarez-Ortega C, Zamora Aunon P, Rodriguez IR, Gomez Prieto P, Buno Soto A, Canales Albendea M, Albaladejo A, Mediavilla G, Feliu Batlle J, Rodriguez Fraga O, Martinez Monzonis A, Gonzalez-Costello J, Serrano Antolin JM, Cadenas Chamorro R, Gonzalez-Juanatey JR, Lopez-Sendon J; CARDIOTOX registry investigators. Cardiovascular risk factors during cancer treatment. Prevalence and prognostic relevance: insights from the CARDIOTOX registry. Eur J Prev Cardiol. 2022 May 6;29(6):859-868. doi: 10.1093/eurjpc/zwaa034. PMID 33624069
- See also: Web site of the study — http://www.cardiotox.org